CLINICAL TRIAL: NCT02722447
Title: Rivaroxaban for the Treatment of Symptomatic Isolated Distal Deep Vein Thrombosis
Acronym: RIDTS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Ageno (Other)
Responsible Party: Sponsor-Investigator, Walter Ageno, Associate Professor of Medicine, Università degli Studi dell'Insubria
Organization: Università degli Studi dell'Insubria (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-000958-36
Record Dates: First submitted 2016-03-13; First posted 2016-03-30 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Active Comparator): Rivaroxaban 20 mg od for 6 weeks after an initial course of rivaroxaban for 6 weeks (15 mg bid for 3 weeks and 20 mg od for 3 weeks)
  Interventions: Drug: rivaroxaban
- Placebo (Experimental): Placebo for 6 weeks after an initial course of rivaroxaban for 6 weeks (15 mg bid for 3 weeks followed by 20 mg od for 3 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rivaroxaban — Rivaroxaban 20 mg for 6 weeks
  Arms: Rivaroxaban
Drug: Placebo — Placebo for 6 weeks
  Arms: Placebo

SUMMARY:
The treatment of isolated distal deep vein thrombosis remains one of the most debated issues in the field of venous thromboembolism and only very few studies have directly addressed the issue of treatment in objectively confirmed isolated distal deep vein thrombosis. Aim of this study is to assess the long-term risk of recurrent venous thrombotic events in patients with a first acute symptomatic isolated distal deep vein thrombosis of the leg treated with a standard (12 weeks) or with a shorter (6 weeks) duration of therapy with rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Objective diagnosis of isolate distal deep vein thrombosis within 72 hours from the evaluation for inclusion in the study and if any type of parenteral treatment was administered at therapeutic doses for 3 days or less (maximum accepted doses of low molecular weight heparin: 6 doses; of fondaparinux: 3 doses).

Exclusion Criteria:

* Age < 18 years
* Any absolute contraindication to anticoagulant treatment
* Pregnancy or breast-feeding
* Presence of active cancer
* Concomitant presence of proximal deep vein thrombosis or pulmonary embolism
* Any concomitant indication for long-term anticoagulant treatment
* Creatinine clearance ≤30 ml/min, according to Cockcroft-Gault equation
* Cirrhosis Child-Pugh score B or C
* Liver disease associated with coagulopathy and high risk of bleeding
* Any other contraindication to rivaroxaban as per local SmPC
* Failure to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrent venous thromboembolism | 24 months
  Recurrent venous thromboembolism defined as new deep vein thrombosis, extension of distal deep vein thrombosis or pulmonary embolism

SECONDARY OUTCOMES:
Rate of major bleeding events | Until 2 days from the last intake of the study drug
Rate of clinically relevant non-major bleeding events | Until 2 days from the last intake of the study drug
Percentage of patients with residual vein occlusion | 3 months and 24 months
Rate of cardiovascular events | 24 months

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - Ospedale di Faenza, Faenza
  - Ospedale di Padova, Padua
  - Ospedale di Pieve di Soligo, Pieve di Soligo
  - Ospedale di Reggio Emilia, Reggio Emilia
  - University of Siena, Siena
  - Ospedale di Circolo, Varese
  - University Of Insubria, Varese

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ageno W, Bertu L, Bucherini E, Camporese G, Dentali F, Iotti M, Lessiani G, Parisi R, Prandoni P, Sartori M, Visona A, Bigagli E, Palareti G; RIDTS study group. Rivaroxaban treatment for six weeks versus three months in patients with symptomatic isolated distal deep vein thrombosis: randomised controlled trial. BMJ. 2022 Nov 23;379:e072623. doi: 10.1136/bmj-2022-072623. PMID 36520715